CLINICAL TRIAL: NCT05270967
Title: Evaluation of Metabolic Changes in FDG PET/CT Imaging After mRNA-based COVID-19 Vaccination
Brief Title: FDG (Fluorodeoxyglucose) Findings After COVID-19 Vaccination
Acronym: fdg
Status: Completed | Type: Observational
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Serkan Isgoren, associate professor of nuclear medicine, Kocaeli University
Other Study IDs: GOKAEK-2021/14.18
Record Dates: First submitted 2022-03-05; First posted 2022-03-08 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-03

CONDITIONS: Vaccine Reaction; Oncology
Keywords: covid-19; vaccine; pet/ct; FDG; mRNA
MeSH Terms: conditions — Neoplasms; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: F-18 FDG PET/CT imaging — Oncological imaging
Biological: Pfizer/biontech mRNA vaccine — COVID-19 vaccine

SUMMARY:
It is important to evaluate the vaccine-related metabolic changes on FDG PET/CT to avoid confusing results. The investigators aimed to assess the frequency and intensity of regional and systemic metabolic PET/CT changes of patients who received the mRNA-based COVID-19 vaccine (BNT162b2-Pfizer/BioNTech) and to analyze possible factors affecting these changes.

ELIGIBILITY:
Inclusion Criteria:

* patients referred for post-vaccination FDG PET/CT imaging

Exclusion Criteria:

* Disseminated metastatic disease, ipsilateral breast cancer or lymphoma that was likely to involve axilla, and patients who had ipsilateral intense axillary uptake or thyroiditis on their prior imaging, were exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: recently vaccinated patients who underwent FDG PET/CT imaging between July 2021 and December 2021, were included in this prospective analysis
Sampling Method: Non-Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2021-07-29 (Actual); Primary Completion 2022-01-10 (Actual); Study Completion 2022-01-10 (Actual)

PRIMARY OUTCOMES:
to assess the frequency of regional and systemic metabolic PET/CT changes of patients who received the mRNA-based COVID-19 vaccine | 5 month
  Frequency of metabolic changes
to assess the FDG intensity of regional and systemic metabolic PET/CT changes of patients who received the mRNA-based COVID-19 vaccine | 5 month
  FDG intensity of metabolic changes

CONTACTS AND LOCATIONS:
Overall Officials: Serkan Isgoren, Ass prof, Study Chair — Kocaeli University School of Medicine
Locations (1):
- Kocaeli University School of Medicine Dep. of Nuclear Medicine, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
study results

REFERENCES:
- [Result] Cohen D, Krauthammer SH, Wolf I, Even-Sapir E. Hypermetabolic lymphadenopathy following administration of BNT162b2 mRNA Covid-19 vaccine: incidence assessed by [18F]FDG PET-CT and relevance to study interpretation. Eur J Nucl Med Mol Imaging. 2021 Jun;48(6):1854-1863. doi: 10.1007/s00259-021-05314-2. Epub 2021 Mar 27. PMID 33774684